CLINICAL TRIAL: NCT02611531
Title: Video vs. TTG Respiratory Inhaler Technique Assessment and InstructioN (V-TRaIN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12-1844
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Module Education (VME) (Experimental): The RE will provide participants with a tablet device and will demonstrate how to access VME and complete the pre/post e-learning assessments. The RE will provide technical support but will neither participate directly in the education nor help with the self-assessments. The participants will first complete the pre-assessment e-learning tool on the tablet. They will then watch the video instruction that will provide a complete demonstration with verbal instructions on correct inhaler technique. Next the participants will complete the post-assessment e-learning tool. Based on participants' performance, they will be directed to further tailored video-instruction. The cycle of self-assessment and video instruction will continue until sufficient mastery has been achieved.
  Interventions: Behavioral: Video Module Education (VME)
- Teach-To-Goal (TTG) (Active Comparator): Participants assigned to the TTG condition will be provided with an intensive, iterative education and evaluation strategy that consists of the following steps.
  Interventions: Behavioral: Teach-To-Goal (TTG)

INTERVENTIONS:
Behavioral: Video Module Education (VME) — Participants will complete inhaler education on a tablet device
  Arms: Video Module Education (VME)
Behavioral: Teach-To-Goal (TTG) — Participants will complete intensive in-person inhaler education
  Arms: Teach-To-Goal (TTG)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two different ways to teach subjects while hospitalized how to use respiratory inhalers and to follow-up after discharge home from the hospital to determine durability of the education.

DETAILED DESCRIPTION:
Asthma and Chronic obstructive pulmonary disease (COPD) results in over a million hospitalizations in the United States annually and COPD is the third leading cause of 30-day re-hospitalizations. Clinical trials have established the efficacy of treatments primarily dispensed via respiratory inhaler devices that reduce morbidity and health care utilization if they are used correctly. Unfortunately, the effectiveness of these medications in real-world settings is limited by the fact that patients often do not use inhalers correctly. Current guidelines recommend assessing and teaching inhaler technique at all health care encounters, including hospitalization. My work has found that over 75% of hospitalized patients in an urban, predominantly underserved population misuse their respiratory inhalers, highlighting a missed opportunity to educate these patients with high potential to benefit. Hospitalization, therefore, provides a potential 'teachable moment' to correct this misuse. My preliminary data indicate that one strategy, in-person teach-to-goal (TTG), is effective in teaching hospitalized patients proper inhaler technique and is more effective than simple verbal instruction.

While TTG is a promising method to improve care for patients who use inhalers, several limitations prevent widespread adoption. First, TTG relies on in-person assessment and education, as well as training and monitoring instructors to ensure fidelity, making it time-consuming and costly. Also, because a single educational session does not ensure long-term retention, post-discharge reinforcement may be needed, which may be impractical with in-person TTG. One potential method to surmount TTG's limitations is use of interactive video module education (VME), a method that has been used for health education in other clinical contexts. Through iterative self-assessments and video-demonstrations on a tablet computer, VME has the potential to be less costly, maintain fidelity, and be more easily extended into the post-discharge setting than in-person TTG. However, certain questions remain about VME. It is unclear whether VME will yield similar results when compared to TTG, or whether patients will have the ability to, and be willing to use, VME in the post-discharge setting. Therefore, before widespread implementation of VME, it is critical to rigorously develop and test VME for inhaler education in the hospital setting. Ultimately, it will also be important to understand patients' ability and willingness to use post-discharge VME for educational reinforcement to allow for this strategy to transition patients across care settings from hospital to home.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Admission to the inpatient medical service and surgical service
3. Physician-diagnosed COPD or asthma. We will enroll patients even if the primary reason for admission is not COPD or asthma (e.g., patients admitted for heart failure, but with a physician diagnosis of COPD are eligible).

Exclusion Criteria:

1. Currently in an intensive care unit
2. Physician declines to provide consent
3. Patient unable to provide consent (e.g., history of cognitive impairment, unable to understand English) or declines to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with metered dose inhaler (MDI) misuse post VME vs. TTG education. This will provide data on the short-term effectiveness of the interventions. | Up to 30 days
  Assess patient's inhaler technique using Inhaler checklists by the trained assessor.

SECONDARY OUTCOMES:
Symptom burden | Up to 30 days
  Symptom burden will be assessed using interviewer-administered surveys
Quality of Life (QOL) | up to 30 days
  Use validated disease specific QOL tools (i.e., asthma or COPD QOL tools)
self-efficacy of inhaler technique | up to 30 days
  Assess patient's confidence in using their inhalers using a Likert scale response to the question "I am confident that I know how to use this respiratory inhaler correctly."
Utilization of health care services (outpatient visits, ED and hospital admissions, deaths) | Up to 30 days
Lung function | Up to 30 days
  Assess patient's lung function via spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Valerie G Press, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Press VG, Arora VM, Kelly CA, Carey KA, White SR, Wan W. Effectiveness of Virtual vs In-Person Inhaler Education for Hospitalized Patients With Obstructive Lung Disease: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jan 3;3(1):e1918205. doi: 10.1001/jamanetworkopen.2019.18205. PMID 31899529